CLINICAL TRIAL: NCT01220674
Title: Pilot Testing a New Computer-based Screening Tool to Detect Cognitive Impairment
Status: Completed | Type: Observational
Sponsor: University of Nebraska (Other)
Collaborators: Massachusetts Institute of Technology (Other); San Mateo Medical Center (Other); VA Northern California Health Care System (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 0491-10-FB
Record Dates: First submitted 2010-10-12; First posted 2010-10-14 (Estimated); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Cognitive Impairment
Keywords: neuropsychological assessment; cognitive impairment; computer-aided diagnostic tool
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Neuropsychological Tests

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- community dwelling older adults, normal controls: men and women 55 years of age or older who are cognitively intact.
  Interventions: Other: cognitive testing
- community dwelling older adults, mild cognitive impairment: men and women 55 years of age or older who have minimal cognitive decline (MMSE 20-24).
  Interventions: Other: cognitive testing

INTERVENTIONS:
Other: cognitive testing — computer-based cognitive assessment

SUMMARY:
A computer-based neuropsychological assessment tool is being developed to help primary care physicians detect neurological and psychiatric disorders. The first version will be tested against current tests to confirm the tool's effectiveness. Data will be collected on how well the tool detects disease, how well patients understand the instructions and enjoy performing the tasks, and if particular trials or stimuli are too difficult or too easy for all subjects. Adjustments can then be made to the assessment tool, if needed. The initial participants will be age fifty-five to seventy-five with early dementias or mild cognitive impairment to reduce variability.

DETAILED DESCRIPTION:
The investigators are developing a computer-based neuropsychological assessment tool to help primary care physicians detect neurological and psychiatric disorders. To confirm the tool's efficacy, the investigators will first test the prototype against established tests. The investigators propose to collect preliminary data on a limited group of subjects and age-matched controls. Collecting data on a limited group of subjects provides early insight into how well the tool detects disease, how well patients understand the instructions and enjoy performing the tasks, and if particular trials or stimuli are too difficult or too easy for all subjects. With this information, the investigators can make adjustments to the tool if needed and collect additional data on revised versions of the tool. The data will be used to establish the validity, reliability and sensitivity of the tool to generate consistent and accurate scores. The investigators will initially focus on a limited age range (age fifty-five to seventy-five) and limited set of diseases (early dementias or mild cognitive impairment) to reduce variability within the patient and control groups and to gain more statistical power with a smaller group of subjects.

ELIGIBILITY:
Inclusion Criteria:

* Any subject with mild impairment from who has already undergone or will soon undergo a full neuropsychological evaluation.
* Subjects with Clinical Dementia Rating Scale CDR of 0.5-1.0 and Mini-Mental Score 20-26 (or MOCA equivalent, borderline/mild dementia) will be eligible for this group.
* Normal controls without exclusion criteria.

Exclusion Criteria:

* Subjects whose impairment is severe enough to limit their ability to perform the computer-based tasks and/or to provide consent.
* Subjects with history of learning disabilities or mental illness including major depression, bipolar disorder, anxiety disorders, and addiction are excluded because these problems can affect cognitive performance.

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Community-dwelling adults without significant cognitive impairment
Sampling Method: Probability Sample
Enrollment: 152 (Actual)
Dates: Start 2010-12-15 (Actual); Primary Completion 2012-10-31 (Actual); Study Completion 2012-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen J Bonasera, MD, PhD, Principal Investigator — University of Nebraska
Locations (1):
- Unversity of Nebraska Medical Center, Omaha, Nebraska, United States